CLINICAL TRIAL: NCT01762293
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter, Phase IIb Study of Famitinib as Third Line Treatment in Patients With Advanced Colorectal Cancer
Brief Title: A Study of Famitinib in Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMTN-IIb-CRC
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2013-01

CONDITIONS: Colorectal Cancer; Colorectal Cancer Metastatic; Colorectal Cancer Recurrent
Keywords: CRC; Famitinib; Phase II; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — famitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Famitinib (Experimental): Famitinib 25 mg qd p.o. and the medication continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Famitinib
- Placebo (Placebo Comparator): Placebo qd p.o., and the medication continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Famitinib — Famitinib 25 mg p.o. qd
  Arms: Famitinib
Other: placebo — p.o. qd
  Arms: Placebo

SUMMARY:
Famitinib is a tyrosin-inhibitor agent targeting at c-Kit, VEGFR2, PDGFR, VEGFR3, Flt1 and Flt3, and it's anti-angiogenesis effect has been viewed in preclinical tests. Phase I study has shown that the toxicity is manageable.

The purpose of this study is to determine whether Famitinib can improve progression free survival compared with placebo in patients with advanced colorectal cancer who failed in previous at least two lines of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologic confirmed recurrent and/or metastatic CRC and previously received at least two lines of standard therapy failure(must include 5-Fu,irinotecan and oxaliplatin)
* At least one measurable lesion, larger than 10 mm in diameter by spiral CT scan(scanning layer ≤ 5 mm )
* age ≥ 18 and ≤ 70
* ECOG 0-1
* Life expectancy of more than 3 months
* More than 4 weeks after operation, chemotherapy, radiotherapy, cytotoxic agents or tyrosine kinase inhibitors
* Signed and dated informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* Before or at the same time any, second malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Prior therapy with tyrosine kinase -inhibitor agent targeting at VEGFR, PDGFR and c-Kit(e.g sorafenib,sunitinib,regorafenib)
* Any factors that influence the usage of oral administration
* Having obvious gastrointestinal hemorrhagic tendency
* Known Spinal Cord compression or diseases of brain or pia mater by CT /MRI screening
* Organ tumor overloading
* Inadequate hepatic, renal, heart, and hematologic functions (hemoglobin ≤ 90g/L, platelets ≤ 100×10^9/L, neutrophils ≤ 1.5×10^9/L, total bilirubin ≥ 1.25×the upper limit of normal(ULN), and serum transaminase ≥ 1.5×ULN (If liver metastases, serum transaminase≥ 2.5×ULN), creatinine clearance rate ≤ 60ml/min, cholesterol ≥ 1.5×ULN and triglyceride≥ 2.5 x ULN, LVEF: < 50%
* Preexisting uncontrolled hypertension defined as more than 140/90 mmHg despite using single medical therapy, more than cla ss I (NCI CTCAE 3.0 ) myocardial ischemia, arrhythmia, or cardiac insufficiency
* urinary protein≥ ++ or 24-hour urinary protein ≥ 1.0 g
* Long-term untreated wounds or fractures
* Blood coagulation abnormal, having hemorrhagic tendency
* Within 1 year before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism, etc.
* Application of anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues; If the prothrombin time international normalized ratio (INR) ≤ 1.5, with the purpose of prevention, the use of small doses of warfarin (1mg orally, once daily) or low-dose aspirin (between 80mg to 100mg daily) is allowed
* Female: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article. Child bearing potential, a negative urine or serum pregnancy test result before initiating Famitinib. Male: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article.
* Preexisting thyroid dysfunction, even using medical therapy, thyroid function cannot maintain in the normal range
* Abuse of psychiatric drugs or dysphrenia
* Less than 4 weeks from the last clinical trial
* Ascites need treatment
* Immunodeficiency: HIV positive, or other acquired immunodeficiency, congenital immunodeficiency, or organ transplantation
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | 3 years

SECONDARY OUTCOMES:
Objective response rate(ORR) | 12 weeks
Disease Control Rate(DCR) | 12 weeks
Overall Survival(OS) | 3 years
Quality of Life | 42-day cycle visit until disease progress
Number of Participants with Adverse Events as a Measure of Safety | 3 years

OTHER OUTCOMES:
body vitals, laboratory parameters | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Lin, M.D, Principal Investigator — Beijing Cancer Hospital, Peking University; Ruihua Xu, M.D, Principal Investigator — Cancer Center, Sun Yet-sen University
Locations (2):
- China (2):
  - Cancer center, Sun Yet-sen University, Guangzhou, Guangdong
  - Beijing Cancer Hospital, Peking University, Beijing

REFERENCES:
- [Derived] Xu RH, Shen L, Wang KM, Wu G, Shi CM, Ding KF, Lin LZ, Wang JW, Xiong JP, Wu CP, Li J, Liu YP, Wang D, Ba Y, Feng JP, Bai YX, Bi JW, Ma LW, Lei J, Yang Q, Yu H. Famitinib versus placebo in the treatment of refractory metastatic colorectal cancer: a multicenter, randomized, double-blinded, placebo-controlled, phase II clinical trial. Chin J Cancer. 2017 Dec 22;36(1):97. doi: 10.1186/s40880-017-0263-y. PMID 29273089